CLINICAL TRIAL: NCT02063698
Title: A Pilot Randomized, Placebo-Controlled Study to Test Auranofin (Ridaura®) to Control the Paclitaxel-Induced Pain Syndrome (PIAPS)
Brief Title: Auranofin in Decreasing Pain in Patients With Paclitaxel-Induced Pain Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC1364; NCI-2014-00165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1364 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Auranofin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (auranofin) (Experimental): Patients receive auranofin PO on day 2.
  Interventions: Drug: auranofin; Other: questionnaire administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO on day 2.
  Interventions: Other: placebo; Other: questionnaire administration

INTERVENTIONS:
Drug: auranofin — Given PO
  Other Names: Ridaura
  Arms: Arm I (auranofin)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies whether auranofin will relieve pain following paclitaxel in patients who have previously experienced paclitaxel-induced pain. Auranofin is a drug given by mouth to treat other diseases such as rheumatoid arthritis, and is being studied to see if it will decrease pain following paclitaxel.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether one dose of auranofin given the day following administration of paclitaxel decreases pain as assessed by daily completion of the Modified Brief Pain Inventory scale for seven days.

SECONDARY OBJECTIVES:

I. Assess whether auranofin is well tolerated in this setting.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive auranofin orally (PO) on day 2.

ARM II: Patients receive placebo PO on day 2.

After completion of study treatment, patients are followed up at 21-28 days.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count (PLT) >= 100,000/mm^3
* Creatinine =< 2 x upper limit of normal (ULN)
* Either serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) or serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 1.5 x ULN
* Total/direct bilirubin =< 1.5 x ULN
* Alkaline phosphatase =< 1.5 x ULN
* Hemoglobin >= 9 mg/dL
* Negative urine or serum pregnancy test performed =< 7 days prior to registration, for women of childbearing potential only
* Previously experienced paclitaxel induced pain during a current or past paclitaxel treatment that the treating healthcare provider thinks is consistent with the paclitaxel-induced acute pain syndrome; note: formal documentation of prior pain is not required
* Scheduled to receive paclitaxel at a dose >= 70 mg/m^2 =< 14 days from randomization
* Ability to complete the questionnaires or to do so with assistance

Exclusion Criteria:

* Pregnant women
* Nursing women
* Any woman of childbearing potential or male partner of a woman of childbearing potential unwilling to employ acceptable contraception throughout the study and for at least 30 days after the last dose of the study drug
* History of gold-induced disorders, including but not limited to, necrotizing enterocolitis, pulmonary fibrosis, exfoliative dermatitis, bone marrow aplasias or other severe hematologic disorders; history of severe allergic or anaphylactic reactions or hypersensitivity to auranofin or other gold compounds
* Currently receiving Dilantin (phenytoin) or auranofin or another gold-containing compound
* Anticipated use of filgrastim (G-CSF) or sargramostim (GM-CSF) within 30 days after receiving auranofin
* Currently receiving immune-modulating therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2015-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2
Not completed — did not complete booklet for days 2-8 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Auranofin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.0) | 57.4 (9.7) | 60.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Count/Percentage of Patients Who Report Having Experienced the Paclitaxel-induced Pain Syndrome (PIAPS) for One Week After Paclitaxel After Enrollment to the Current Trial, Assessed by the Modified Brief Pain Inventory Scale (BPI)
Description: The primary endpoint is the per arm count/percentage of patients who report having experienced the PIAPS for one week after paclitaxel after enrollment to the current trial. Pain was assessed on the question 'Please rate your pain by circling the one number that best describes your pain at its worst in the last 24 hours'. The count of participants who report having experienced the PIAPS for one week after paclitaxel after enrollment to the current trial circling 'less than 4' and 'greater than or equal to 4' for each day between day 2 to day 8 are reported below. Modified Brief Pain Inventory (BPI) ranges from 0 to 10, with higher scores corresponding to more /worse pain. Fisher's Exact Test will be used to compare the frequency of patients who experienced PIAPS between the two arms.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 14 | 13
Participants
  Day 2: BPI Worst Pain Past 24 Hours: <4 | 10 | 10
  Day 2: BPI Worst Pain Past 24 Hours: >=4 | 4 | 3
  Day 3: BPI Worst Pain Past 24 Hours: <4 | 5 | 7
  Day 3: BPI Worst Pain Past 24 Hours: >=4 | 9 | 6
  Day 4: BPI Worst Pain Past 24 Hours: <4 | 2 | 4
  Day 4: BPI Worst Pain Past 24 Hours: >=4 | 12 | 9
  Day 5: BPI Worst Pain Past 24 Hours: <4 | 3 | 7
  Day 5: BPI Worst Pain Past 24 Hours: >=4 | 11 | 6
  Day 6: BPI Worst Pain Past 24 Hours: <4 | 7 | 8
  Day 6: BPI Worst Pain Past 24 Hours: >=4 | 7 | 5
  Day 7: BPI Worst Pain Past 24 Hours: <4 | 8 | 8
  Day 7: BPI Worst Pain Past 24 Hours: >=4 | 6 | 5
  Day 8: BPI Worst Pain Past 24 Hours: <4 | 10 | 7
  Day 8: BPI Worst Pain Past 24 Hours: >=4 | 4 | 6
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 2: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 1.0, Fisher Exact
Statistical Analysis 2: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 3: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 0.45, Fisher Exact
Statistical Analysis 3: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 4: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 0.38, Fisher Exact
Statistical Analysis 4: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 5: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 0.12, Fisher Exact
Statistical Analysis 5: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 6: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 0.70, Fisher Exact
Statistical Analysis 6: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 7: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 1.0, Fisher Exact
Statistical Analysis 7: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Day 8: BPI Worst Pain Past 24 Hours; Test type: Superiority; p = 0.44, Fisher Exact

2. Primary Outcome: Area Under the Curve (AUC) Summary of Worst Pain in the Last 24 Hours From Days 2 to 8
Description: Area under the curve (AUC) Summary of Worst Pain in the last 24 hours from days 2 to 8. On a scale of 0-100, with 100=Best QOL. Pain was assessed on the question 'Please rate your pain by circling the one number that best describes your pain at its worst in the last 24 hours.' Modified Brief Pain Inventory (BPI) ranges from 0 to 10, with higher scores corresponding to more pain. The AUC for this question was then calculated and ranged from 0-100, with higher scores corresponding to less/improved pain. The Equal Variance T-test will be used to compare the average AUC for worst pain between the two arms.
Time Frame: Up to 8 days
Measure: Mean (Standard Deviation); unit: score on a scale * day
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 14 | 12
score on a scale * day | 55.1 (19.0) | 61.3 (21.8)
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.44, Equal variance t-test

3. Secondary Outcome: Normalized AUC for BPI Average Pain From the Modified BPI in the Last 24 Hours From Days 2 to 8
Description: Normalized AUC for BPI Average pain from the modified BPI in the last 24 hours from days 2 to 8. On a scale of 0-100 with 100:Best QOL. Pain was assessed on the question 'Please rate your pain by circling the one number that best describes your pain on the average.' Modified Brief Pain Inventory (BPI) ranges from 0 to 10, with higher scores corresponding to more pain. The AUC for this question was then calculated and ranged from 0-100, with higher scores corresponding to less/improved pain. The Equal Variance T-test will be used to compare the average AUC for worst pain between the two arms.
Time Frame: Up to 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
score on a scale | 67.0 (17.9) | 78.1 (18.2)
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.13, Equal variance t-test

4. Secondary Outcome: Worst Toxicity Assessed Using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4
Description: The maximum grade for each type of toxicity will be recorded for each patient. The count of participants with worst adverse events considered at least possibly related to treatment by maximum grade are reported below.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
Participants
  1-Mild | 9 | 7
  2-Moderate | 4 | 1
  3-Severe | 2 | 6
  4-Life-Threatening | 0 | 1

5. Secondary Outcome: Cramp Pain as Measured by the Paclitaxel-Induced Acute Pain Syndrome (PIAPS) Symptom Summary on Day 5
Description: Cramp Pain as measured by the Paclitaxel-Induced Acute Pain Syndrome (PIAPS) Symptom Summary on Day 5. The PIAPS question 'Please place a check mark (√) by all appropriate words that could be used to describe any pain you have had in the last 24 hours'. The number of participants who completed this question on day 5 were analyzed (those who checked 'cramping' are summarized by the 'Yes' row below and those who did not check 'cramping' are summarized by the 'No' row below. Those who did not complete the symptom summary are summarized by the 'Missing' row.) The chi-square test was used.
Time Frame: Up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
Participants
  Missing | 1 | 2
  No | 14 | 9
  Yes | 0 | 4
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.025, Chi-squared

6. Secondary Outcome: Gnawing Pain as Measure by the Paclitaxel-Induced Acute Pain Syndrome (PIAPS) Symptom Summary on Day 8
Description: Gnawing Pain as measured by the Paclitaxel-Induced Acute Pain Syndrome (PIAPS) Symptom Summary on Day 8. The PIAPS question 'Please place a check mark (√) by all appropriate words that could be used to describe any pain you have had in the last 24 hours'. The number of participants who completed this question on day 8 were analyzed (those who checked 'gnawing' are summarized by the 'Yes' row below and those who did not check 'gnawing' are summarized by the 'No' row below. Those who did not complete the symptom summary are summarized by the 'Missing' row.) The chi-square test was used.
Time Frame: Up to 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
Participants
  Missing | 1 | 2
  No | 14 | 8
  Yes | 0 | 5
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.01, Chi-squared

7. Secondary Outcome: Location of New Pain Patient Had in the Last 24 Hours on Day 5 PIAPS Upper Arm Pain
Description: Location of New Pain Patient had in the last 24 hours on day 5 PIAPS Upper arm pain. PIAPS question: "Please indicate where any new pains are/were located by placing a check mark (√) next to the location. Please mark all that apply:" The number of participants who completed this question on day 5 were analyzed (those who checked 'arm, above the elbow' are summarized by the 'Yes' row below and those who did not check 'arm, above the elbow' are summarized by the 'No' row below. Those who did not complete the symptom summary are summarized by the 'Missing' row.) The chi-square test was used.
Time Frame: Up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
Participants
  Missing | 1 | 2
  No | 9 | 13
  Yes | 5 | 0
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.02, Chi-squared

8. Secondary Outcome: Location of New Pain Patient Had in the Last 24 Hours on Day 5 PIAPS Lower Arm Pain.
Description: Location of New Pain Patient had in the last 24 hours on day 5 PIAPS Lower arm pain. PIAPS question: "Please indicate where any new pains are/were located by placing a check mark (√) next to the location. Please mark all that apply:" The number of participants who completed this question on day 5 were analyzed (those who checked 'arm, between the elbows and wrists' are summarized by the 'Yes' row below and those who did not check 'arm, between the elbows and wrists' are summarized by the 'No' row below. Those who did not complete the symptom summary are summarized by the 'Missing' row.) The chi-square test was used.
Time Frame: Up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
Participants
  Missing | 1 | 2
  No | 8 | 13
  Yes | 6 | 0
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.01, Chi-squared

9. Secondary Outcome: Location of New Pain Patient Had in the Last 24 Hours on Day 6 PIAPS Lower Arm Pain.
Description: Location of New Pain Patient had in the last 24 hours on day 6 PIAPS Lower arm pain. PIAPS question: "Please indicate where any new pains are/were located by placing a check mark (√) next to the location. Please mark all that apply:" The number of participants who completed this question on day 5 were analyzed (those who checked 'arm, between the elbows and wrists' are summarized by the 'Yes' row below and those who did not check 'arm, between the elbows and wrists' are summarized by the 'No' row below. Those who did not complete the symptom summary are summarized by the 'Missing' row.) The chi-square test was used.
Time Frame: Up to 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 15
Participants
  Missing | 1 | 2
  No | 10 | 13
  Yes | 4 | 0
Statistical Analysis 1: Comparison: Arm I (Auranofin) vs Arm II (Placebo); Test type: Superiority; p = 0.04, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed the study. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm I (Auranofin) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 5/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Auranofin) (N=15) | Arm II (Placebo) (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Auranofin) (N=15) | Arm II (Placebo) (N=15)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 14 (14) | 15 (15)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes